CLINICAL TRIAL: NCT05036759
Title: 68Ga-FAPI PET/MR for Intracranial and Carotid Atherosclerosis
Brief Title: 68Ga-FAPI PET/MR for Atherosclerosis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-FAPI-PET/MR
Record Dates: First submitted 2021-08-30; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; 68Ga-FAPI; PET/MR
MeSH Terms: conditions — Atherosclerosis | interventions — 68Ga-FAPI

STUDY DESIGN:
Intervention Model Description: 68Ga-FAPI PET/MR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI, PET/MR (Experimental): inject 68Ga-FAPI，and then perform PET/MR
  Interventions: Drug: 68Ga-FAPI

INTERVENTIONS:
Drug: 68Ga-FAPI — intravenously injected with 68Ga-FAPI
  Other Names: 68Ga-fibroblast activating protein inhibitors

SUMMARY:
A thin-cap fibroatheroma with a large necrotic core and macrophage infiltration marks the vulnerable plaque. Fibroblast activating protein (FAP) is an active serine protease, which can degrade type I collagen, potentially thinning the fibrous cap. Thus we speculate that atherosclerotic plaque could be imaged with 68Ga-FAPI PET/MR.

DETAILED DESCRIPTION:
A thin-cap fibroatheroma with a large necrotic core and macrophage infiltration marks the vulnerable plaque. Fibroblast activating protein (FAP) is an active serine protease, which can degrade type I collagen, potentially thinning the fibrous cap. Previous ex vivo analysis of human aortic atheromata revealed that FAP was expressed in atherosclerotic plaques, and higher FAP expression was detected in thin fibrous caps than thick caps. Constitutive Fap deletion in atherosclerosis-prone mice models could reduce plaque formation and improve plaque stability with increased fibrous cap thickness. Thus we speculate that atherosclerotic plaque could be imaged with 68Ga-FAPI PET/MR.

ELIGIBILITY:
Inclusion Criteria:

* intracranial or carotid atherosclerosis patients
* signed informed consent

Exclusion Criteria:

* pregnancy, breastfeeding
* contradictions of MRI
* unstable vital signs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | through study completion, an average of 2 years
  Diagnostic performance of 68Ga-FAPI PET/MR for intracranial or carotid atherosclerosis

SECONDARY OUTCOMES:
SUVmax | through study completion, an average of 2 years
  The difference of SUVmax between asymptomatic and symptomatic atherosclerotic patients
FAPI expression | through study completion, an average of 2 years
  The correlation of SUVmax and pathological FAPI expression

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Yang, M.D., Principal Investigator — Peking Union Medical College Hospital; Meiqi Wu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No